CLINICAL TRIAL: NCT03775668
Title: A Phase 1, Open-Label, Single-Dose Study to Assess the Mass Balance, Pharmacokinetics and Metabolism of Intravenously Administered 14C-AAI101 in Healthy Male Subjects
Brief Title: Single Dose Mass Balance Study With C14 - Labeled AAI101 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allecra (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-104
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — enmetazobactam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 µCi of 14C-AAI101 + 500 mg AAI101 (Experimental): 14C-AAI101 + 500 mg AAI101 iv infusion
  Interventions: Drug: 1 µCi of 14C-AAI101 + 500 mg AAI101

INTERVENTIONS:
Drug: 1 µCi of 14C-AAI101 + 500 mg AAI101 — Single dose open label
  Other Names: 14C-AAI101 + 500 mg AAI101 iv infusion

SUMMARY:
This is an open-label, single dose, pharmacokinetic (PK) study conducted at 1 study center in the United States (USA). This study will evaluate the absorption, distribution, metabolism, and elimination (ADME), mass balance, safety, and tolerability of a single dose of intravenously administered 14C-AAI101.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willing to sign the Informed Consent Form (ICF)
2. BMI 18.0 - 35.0 kg/m2, inclusive,
3. Subjects with normal renal function as evidenced by creatinine clearance (CLcr).
4. Judged to be in good health in the opinion of the Investigator on the basis of a medical evaluation that reveals the absence of any clinically significant abnormality
5. Content of 14C in one or both (at Investigator's discretion) of urine and blood (or plasma) samples obtained at Screening does not significantly exceed the general environmental background 14C level.

Exclusion Criteria:

1. Clinically significant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at Screening, Day -1 or pre-dose on Day 1 that the Investigator judges may put at risk achieving the objectives of the trial or protecting the safety of the volunteer.
2. Documented congenital or acquired long QT syndrome.
3. Corrected QT interval (QTc) using Fridericia correction (QTcF) at Screening or pre dose (Day 1) >450 ms.
4. Family history of long QT syndrome or of unexplained sudden death in a first-degree relative under age 50.
5. History of multiple and/or severe allergies to drugs or foods or a history of anaphylactic reaction.
6. History of cancer judged not to be in full remission for at least 5 years (except basal cell skin cancer or squamous cell skin cancer with history of curative treatment and no recurrence for at least 1 year), as judged by the Investigator.
7. History of active alcoholism or drug abuse within the last 2 years prior to study drug administration. Acceptable use history is typical consumption of up to 14 units per week (1 unit equals 250 mL beer, 75 mL wine, 25 mL spirits per week), or per judgment of the Investigator.
8. Regular alcohol consumption in males >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type).
9. Recent history of incomplete bladder emptying with voiding or of awaking more than once at night to void.
10. Usual habit of less than one or more than three bowel movements per day.
11. Acute illness within 14 days prior to study drug administration unless mild in severity and enrollment is approved by both Investigator and Sponsor's medical representative.
12. Presence of active infection requiring antibiotic treatment.
13. Concomitant or prior use (within 60 days prior to study drug administration) of medications known to affect the elimination of serum creatinine (e.g., trimethoprim or cimetidine) or to compete for renal tubular secretion (e.g., probenecid).
14. Allergy, hypersensitivity or intolerance to β-lactam antibiotics and/or cephalosporin-class antibiotics in the medical history.
15. Current smokers and those who have smoked within the last 12 months; this includes cigarettes, e-cigarettes and nicotine replacement or nicotine containing products.
16. Participation in another investigational drug trial within 30 days prior to study drug administration (or 5 times the half-life of the drug, whichever is longer) or exposure to more than three new investigational agents within 12 months prior to study drug administration.
17. Exposure to radiation for therapeutic or diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton) within the last 12 months prior to dosing of the investigational drug, or an occupationally exposed worker
18. Participation in another clinical trial in which a [14C]-labeled drug was administered within the year prior to Day -1.
19. Donation or loss of more than 450 mL blood during the 3 months before the start of and during Screening.
20. Serum Alkaline phosphatase (AP) > 1.5x upper limit of normal (ULN).
21. Serum transaminase [alanine aminotransferase (ALT) or aspartate aminotransferase (AST)] > ULN.
22. Serum uric acid > ULN.
23. Positive serology for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti HCV) or human immunodeficiency virus antibodies (anti-HIV)-1/2 at Screening.
24. Positive urine screen of drugs of abuse or alcohol breath test at Screening and/or Day 1.
25. Strenuous or unaccustomed activity, sunbathing, or contact sports within 96 hours (4 days) prior to entry in the clinic research center.
26. Legal incapacity or limited legal capacity.
27. Any clinically significant medical condition, i.e., one which in the opinion of the Investigator would increase risk to the subject's health if participating in this study or would increase risk of not achieving the study objectives.
28. Use of any prescription or non-prescription drugs, including over-the-counter medication, non-routine vitamins and herbal products within 2 weeks prior to study drug administration unless discussed and agreed with the Sponsor's medical representative in writing.

    -

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Concentrations of total radiolabelled 14C-content in blood, plasma, urine, and feces. | Up to 7 days post dosing
Concentration of parent AAI101 in plasma and urine. | Up to 7 days post dosing

SECONDARY OUTCOMES:
Metabolite profiling for pooled plasma, urine and feces If > 10% of total radioactivity is recovered in the respective excreta sample/collection. | Up to 7 days post dosing
Calculation of cumulative urinary and fecal recovery of total radioactivity, and calculation of mass balance as a sum of the percentages of total radioactivity recovered in urine and feces. | Up to 7 days post dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron Clinical Pharmacology Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No